CLINICAL TRIAL: NCT03670017
Title: GIDE - Glucose Time-In-Range Development Evaluation
Brief Title: Glucose Time-In-Range Development Evaluation
Acronym: GIDE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of Funding
Sponsor: Washington University School of Medicine (Other)
Collaborators: OptiScan Biomedical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GIDE Study
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Results first posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: ICU; Dysglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Time In Range during OptiScanner Connection (Other): Participants will be connected to the OptiScanner 5000 for up to 72 hours.
  Interventions: Device: OptiScanner® 5000 Glucose Monitoring System

INTERVENTIONS:
Device: OptiScanner® 5000 Glucose Monitoring System — The study population includes surgical critical care patients who require blood glucose monitoring. Subjects must have a vascular access device [i.e., Central Venous Catheters (CVC), Multi-lumen Access Catheters (MAC) either in place or to be placed with an expected usage of at least 48 hours. During Phase One of the trial, patients will be connected to the OptiScanner for up to 72 hours and the hospital's current standard of care for glucose management will be followed.

SUMMARY:
The study will evaluate patients requiring frequent glucose monitoring in a Surgical ICU. The study population includes surgical critical care patients who require blood glucose monitoring. Subjects must have a vascular access device [i.e., Central Venous Catheters (CVC), Multi-lumen Access Catheters (MAC) either in place or to be placed with an expected usage of at least 48 hours. During Phase One of the trial, patients will be connected to the OptiScanner for up to 72 hours and the hospital's current standard of care for glucose management will be followed.

DETAILED DESCRIPTION:
Hyperglycemia, hypoglycemia and glycemic variability are independently associated with morbidity and mortality of critically ill patients. Blood glucose control with insulin has the potential to decrease morbidity and mortality of intensive care unit (ICU) patients. Blood glucose control with insulin, however, is associated with an increased risk of hypoglycemia and may not decrease glycemic variability. In addition, blood glucose control with insulin utilizing manual systems for glucose measurement is blood-consuming and time-consuming, since frequent blood draws for glucose measurements are necessary in order to achieve blood glucose control.

Automated, frequent, plasma-based glucose monitoring with the OptiScanner 5000 glucose monitoring system has the potential to improve a patient's glucose TIR by improving all 3 domains of glycemic control: reducing hyperglycemia while at the same time preventing hypoglycemia and reducing glycemic variability. Second, it could reduce the workloads associated with the high number of blood samples to be obtained and analyzed.

The primary objective of this study is to observe the Time-in-Range for patients whose glycemic control is being monitored with the OptiScanner system. A secondary objective is assessment of the time it takes the patient to achieve in range glucose values while connected to the OptiScanner. The study will evaluate patients requiring frequent glucose monitoring in a Surgical ICU.

The study population includes surgical critical care patients who require blood glucose monitoring. Subjects must have a vascular access device [i.e., Central Venous Catheters (CVC), Multi-lumen Access Catheters (MAC) either in place or to be placed with an expected usage of at least 48 hours. During Phase One of the trial, patients will be connected to the OptiScanner for up to 72 hours and the hospital's current standard of care for glucose management will be followed. Currently glucose values are measured using point of care glucose meters and/or by collecting a blood sample and sending it to the hospital laboratory. Patients' glucose values are currently monitored depending on their clinical condition with the frequency of glucose measurement typically occurring every one to four hours. Patients enrolled in this study will still be monitored in this same manner, depending on their clinical condition (using point of care meters and/or blood collection for the lab). The additional continuous monitoring provided by the OptiScanner may introduce additional glucose measurements. The clinical care team will be advised to confirm any OptiScanner glucose value (using routine clinical care methods) before making any modifications to the patient's clinical care based on the OptiScanner result (i.e. increase, decrease, stop insulin drip, etc.). A research team member will be at the bedside during the patients' connection to the OptiScanner to ensure that the clinical team does not use the OptiScanner results to direct patient care and to observe the overall clinical care glucose management of the patient. Clinical data will be captured on the participants.

ELIGIBILITY:
Inclusion Criteria

1. Signed informed consent by the participant or his/her legally authorized representative;
2. At least 18 years old;
3. Admitted to a Surgical Intensive Care Unit (SICU) or planned admission to a Surgical ICU at time of screening
4. Expected SICU stay of at least 48 hours at the time of enrollment
5. A vascular access device available for connection to the OptiScanner is either already in-place, or is planned to be placed with an expected usage of at least 48 hours.

Exclusion Criteria

1. Positive Human chorionic gonadotropin (HcG) (serum or urine ) in women of childbearing potential (age < 60) who are not known to be surgically sterile and those that are obviously pregnant.
2. Patients undergoing peritoneal dialysis within the past week.
3. Patients actively receiving intravenous immunoglobulin therapy.
4. Patients receiving intravenous administration of high dose ascorbate (IVC) for the treatment of patients with cancer.
5. Patients following the administration of a D-Xylose absorption test < 12 hours
6. Patients being treated with Sodium Thiosulfate
7. Patients being receiving IV glycerol
8. Patients receiving substances containing maltose, or substances that can be metabolized into maltose. These substances include Extraneal, Gamimune N, HepaGam B, Octagam, Vaccinia Immune Globulin, and WinRho SDF Liquid.
9. Hct <15% within 24 hours of screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Bochicchio, MD MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Time In Range During OptiScanner Connection
Started | 68
Completed | 50
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | Time In Range During OptiScanner Connection
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 41
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Glucose Time-in-range (TIR)
Description: Glucose time in range will be defined by participant's clinical care defined target glucose range
Time Frame: Up to 72 hours
Population: The percentage of time in range is all that is available. The company declared bankruptcy due to COVID 19. Raw data is no longer available.
Measure: Number; unit: percentage of time in range
Arm/Group | Time In Range During OptiScanner Connection
Number analyzed (Participants) | 50
percentage of time in range | 55

2. Secondary Outcome: Assessment of the Time it Takes the Patient to Achieve in Range Glucose Values While Connected to the OptiScanner.
Description: Evaluation of the amount of time required for a patient to have in range glucose values
Time Frame: Up to 72 hours
Population: The sponsor went out of business prior to completing the analysis for this endpoint therefore the information is not available.
Arm/Group | Time In Range During OptiScanner Connection
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Time In Range During OptiScanner Connection
All-Cause Mortality (participants affected / at risk) | 6/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT03670017/Prot_000.pdf